CLINICAL TRIAL: NCT04788459
Title: A Phase I/II Study to Assess the Safety and Immunogenicity of COVID-eVax, a Candidate Plasmid DNA Vaccine for COVID-19, in Healthy Adult Volunteers
Brief Title: Safety and Immunogenicity of COVID-eVax, a Candidate Plasmid DNA Vaccine for COVID-19, in Healthy Adult Volunteers
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The good progress of the Italian national vaccination campaign against COVID-19 made impossible to complete the study as planned.
Sponsor: Takis (Industry)
Collaborators: Rottapharm Biotech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: COV-1/2-01; 2020-003734-20 (EudraCT Number)
Record Dates: First submitted 2021-03-01; First posted 2021-03-09 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2021-12

CONDITIONS: COVID-19; Protection Against COVID-19 and Infections With SARS-CoV- 2; COVID-19 Immunisation
Keywords: Infections Viral; Coronavirus Disease 2019; Respiratory Tract Infections; Vaccine; SARS-COV-2
MeSH Terms: conditions — COVID-19; Virus Diseases; Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 0.5 mg PB (Experimental): 0.5 mg PB (Prime-Boost, 4 weeks apart) - Total dose: 1 mg
  IM injection + electroporation by IGEA Cliniporator® and EPSGun, on Day 1 and Day 29
  Interventions: Biological: COVID-eVax; Device: Cliniporator® and EPSGun
- 1 mg PB (Experimental): 1 mg PB (Prime-Boost, 4 weeks apart) - Total dose: 2 mg
  IM injection + electroporation by IGEA Cliniporator® and EPSGun, on Day 1 and Day 29
  Interventions: Biological: COVID-eVax; Device: Cliniporator® and EPSGun
- 2 mg PB (Experimental): 2 mg PB (Prime-Boost, 4 weeks apart) - Total dose: 4 mg
  IM injection + electroporation by IGEA Cliniporator® and EPSGun, on Day 1 and Day 29
  Interventions: Biological: COVID-eVax; Device: Cliniporator® and EPSGun
- 2 mg P (Experimental): 2 mg P (Prime) - Total dose: 2 mg
  IM injection + electroporation by IGEA Cliniporator® and EPSGun, on Day 1
  Interventions: Biological: COVID-eVax; Device: Cliniporator® and EPSGun

INTERVENTIONS:
Biological: COVID-eVax — Plasmid DNA Vaccine for COVID-19
Device: Cliniporator® and EPSGun — IGEA Electroporation Device

SUMMARY:
This is a multicentre, open-label Phase 1/2 study, with a first-in-human (FIH) dose escalation part (Phase 1 study) followed by an open-label single arm (or two-arms, randomized) dose expansion part (Phase 2 study). The vaccine will be administered by intramuscular (IM) injection followed by electroporation (EP) applied to the injection site.

The study is aimed at assessing the safety and immunogenicity of COVID-eVax, a DNA plasmid-based vaccine whose target antigen is a portion of the S protein of SARS-CoV-2 virus (the Receptor Binding Domain located in the CTD1 of the S1 region of the S protein).

In animal models COVID-eVax was safe and induced high immunological humoral and cellular response.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent obtained before undergoing any study-specific procedure
2. Healthy male or female aged ≥18 and ≤ 65 years
3. Body Mass Index >18.5 and ≤30 kg/m2
4. Vital signs within the following values or ranges:

   1. Body temperature ≤ 37,5 °C
   2. Pulse frequency ≥51 and ≤100 beats per minute
   3. Diastolic BP ≥60 mmHg, ≤ 90 mmHg
   4. Systolic BP ≥ 90 mmHg, ≤ 140 mmHg
   5. Respiratory rate ≥ 12 breaths per minute, ≤ 16 breaths per minute
5. ECG at screening normal or with no clinically significant findings (pre-excitation syndromes, e.g., Wolff-Parkinson-White syndrome are absolute exclusion criteria)
6. Laboratory examinations within normal reference range or with no clinically significant abnormalities
7. Absence of any respiratory and flu-like symptoms
8. Non-pregnant women of childbearing potential, willing to practice a highly effective method of contraception from enrolment up to study completion or at least 90 days after the last vaccination in case of withdrawal
9. For sexually active men with a female partner of childbearing potential, willingness to use a condom and to refrain from donating sperm from enrolment up to study completion or at least 90 days after the last vaccination in case of withdrawal
10. Agreement to refrain from blood donation during the course of the study
11. Able and willing to comply with all study procedures.

Exclusion Criteria:

1. History of confirmed infection with SARS-CoV-2, by positive nasopharyngeal swab or by positive serological test for SARS-CoV-2 antibodies
2. Positive serological test for SARS-CoV-2 antibodies at screening
3. Subjects at high risk of SARS-CoV-2 infection prior or during the trial, including:

   1. subjects with any known exposure in the 4 weeks before enrolment
   2. close contacts of suspected or confirmed COVID-19 or SARS-CoV-2 infection cases
   3. subjects quarantined for any reason
   4. frontline healthcare professionals working in Emergency departments, ICU and other higher risk healthcare areas
4. Positive serological tests for:

   1. Hepatitis B surface antigen (HBsAg)
   2. Hepatitis C antibodies
   3. Human Immunodeficiency Virus (HIV) antibodies
5. Subjects with any of the following specific contraindications, even in medical history:

   1. Type 2 diabetes or glucose intolerance, even if controlled
   2. Hypertension, even if controlled
   3. chronic obstructive pulmonary disease (COPD)
   4. Any cardiac disease, even if not evident at ECG
   5. Pacemaker
6. Use of any investigational drugs/treatments, or enrolment in a clinical trial during the 6 months preceding screening
7. Prior administration of any vaccine in the 2 weeks preceding screening
8. Administration of any monoclonal or polyclonal antibody product within 4 weeks preceding screening
9. Administration of any blood product within 3 months of screening
10. Current or prior administration, within the 6 months preceding screening, of immunosuppressants (inhaled, topical skin and/or eye drop-containing corticosteroids; a short course of corticosteroids, defined as ≤20 mg/day prednisone or equivalent for 10 days, and low-dose methotrexate are allowed until 4 weeks prior to screening)
11. Any prior major surgery or any chemo- or radiation therapy within 5 years of screening
12. Current or suspected immunosuppressive or immunodeficient state, including HIV infection, asplenia, recurrent severe infections
13. Active, known, or suspected autoimmune disease (except mild psoriasis, well-controlled autoimmune thyroid disease, vitiligo or stable coeliac disease not requiring immunosuppressive or immunomodulatory therapy)
14. Bleeding disorders (e.g. coagulopathy or platelet disorder or coagulation factor deficiency) or prior history of significant bleeding or bruising following IM injections or venipuncture
15. History of seizures or mental illness
16. History of allergy to vaccines or of severe allergic reaction of any kind
17. Metal implants within 20 cm of the planned site(s) of injection
18. Presence of keloid scar formation or hypertrophic scar, or other clinically significant medical condition at the planned site(s) of injection
19. Any abnormality or permanent body art (e.g. tattoos) that would interfere with the ability to observe local reactions at the injection site in the deltoid area
20. History of alcohol or drug abuse during the 12 months preceding the screening
21. Pregnancy (i.e. positive pregnancy test) or willingness/intention to become pregnant during the study
22. Breastfeeding
23. Any other clinically relevant disease and condition that, in the opinion of the Investigator, may jeopardize efficacy or safety assessments or may compromise the subject's safety during trial participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
Incidence of solicited local Adverse events (AEs) at the injection site (for Phase 1) | Through 7 days post-each vaccination
Incidence of solicited systemic AEs (for Phase 1) | Through 7 days post-each vaccination
Incidence of unsolicited AEs (for Phase 1) | through 4 weeks post-each vaccination
White Blood Cell (WBC) levels (for Phase 1) | through 4 weeks post-each vaccination
  Change from baseline at specific timepoints
Red Blood Cell (RBC) levels (for Phase 1) | through 4 weeks post-each vaccination
  Change from baseline at specific timepoints
Platelets levels (for Phase 1) | through 4 weeks post-each vaccination
  Change from baseline at specific timepoints
Alanine Transaminase (ALT) levels (for Phase 1) | through 4 weeks post-each vaccination
  Change from baseline at specific timepoints
Aspartate Transaminase (AST) levels (for Phase 1) | through 4 weeks post-each vaccination
  Change from baseline at specific timepoints
Creatine Phosphokinase (CPK) levels (for Phase 1) | through 4 weeks post-each vaccination
  Change from baseline at specific timepoints
Quantitative antibody titers, binding to the specific SARS-CoV-2 antigen (for Phase 2) | through 4 weeks post-last vaccination
  Geometric Mean Titer (GMT) and Geometric Mean Fold Rise (GMFR) from baseline
SARS-CoV-2 neutralizing antibody titer (for Phase 2) | through 4 weeks post-last vaccination
  GMT and GMFR from baseline
Change from baseline in antigen-specific cellular immune responses to SARS-CoV-2 (for Phase 2) | through 4 weeks post-last vaccination
  Interferon-gamma (IFN-γ) ELISpot
Percentage of subjects who seroconverted (for Phase 2) | through 4 weeks post-last vaccination

SECONDARY OUTCOMES:
Quantitative antibody titers, binding to the specific SARS-CoV-2 antigen (for Phase 1) | through 4 weeks post-last vaccination
  GMT and GMFR from baseline
SARS-CoV-2 neutralizing antibody titer (for Phase 1) | through 4 weeks post-last vaccination
  GMT and GMFR from baseline
Change from baseline in antigen-specific cellular immune responses to SARS-CoV-2 (for Phase 1) | through 4 weeks post-last vaccination
  Interferon-gamma (IFN-γ) ELISpot
Percentage of subjects who seroconverted (for Phase 1) | through 4 weeks post-last vaccination
Incidence of unsolicited AEs (for Phase 1) | through study completion (6 months)
Incidence of solicited local AEs at the injection site (for Phase 2) | Through 7 days post-each vaccination
Incidence of solicited systemic AEs (for Phase 2) | Through 7 days post-each vaccination
Incidence of unsolicited AEs (for Phase 2) | through 4 weeks post-each vaccination
White Blood Cell (WBC) levels (for Phase 2) | through 4 weeks post-each vaccination
  Change from baseline at specific timepoints
Red Blood Cell (RBC) levels (for Phase 2) | through 4 weeks post-each vaccination
  Change from baseline at specific timepoints
Platelets levels (for Phase 2) | through 4 weeks post-each vaccination
  Change from baseline at specific timepoints
Alanine Transaminase (ALT) levels (for Phase 2) | through 4 weeks post-each vaccination
  Change from baseline at specific timepoints
Aspartate Transaminase (AST) levels (for Phase 2) | through 4 weeks post-each vaccination
  Change from baseline at specific timepoints
Creatine Phosphokinase (CPK) levels (for Phase 2) | through 4 weeks post-each vaccination
  Change from baseline at specific timepoints
Incidence of unsolicited AEs (for Phase 2) | through study completion (6 months)

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - San Gerardo Hospital, Monza
  - Istituto Nazionale Tumori, IRCCS, Fondazione G. Pascale, Naples
  - INMI Lazzaro Spallanzani, Rome
  - - CRC Centro Ricerche Cliniche di Verona, Verona